CLINICAL TRIAL: NCT07253987
Title: Cancer Survivors Program: Effectiveness of Monitoring Adverse Events After Completion of Curative Treatment for Breast and Prostate Cancer
Brief Title: Cancer Survivors Program
Acronym: SURV-QoL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masaryk Memorial Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: A8/25_SURV-QoL; A8/25 (Other: Masaryk Memorial Cancer Institute)
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer Patients; Breast Cancer Patients
Keywords: cancer survivors; breast cancer; prostate cancer; neo-/adjuvant chemotherapy; quality of life
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): screening of adverse effects of curative therapy + quality of life screening
  Interventions: Other: active screening of adverse effects of anticancer therapy based on specific questionnaire + quality of life screening
- Control (No Intervention): quality of life screening

INTERVENTIONS:
Other: active screening of adverse effects of anticancer therapy based on specific questionnaire + quality of life screening — Based on the Questionnaire for the Assessment of Difficulties after the completion of cancer treatment, the attending physician will assess the need for intervention and respond appropriately to the reported problems. Intervention is assessed as education by the physician, the use of medication, or referral of the patient to a specialized outpatient clinic.
  Arms: Interventional

SUMMARY:
The questionnaire for assessment of adverse events after completion of cancer treatment, which is being piloted at the Masaryk Memorial Cancer Institute, aims to detect a wide range of adverse effects early on, thus facilitating adequate intervention and planning of follow-up care for all cancer survivors.

DETAILED DESCRIPTION:
According to the current recommendations of the European Society for Medical Oncology (ESMO), comprehensive care for cancer survivors should focus on five main areas: 1) the physical effects of the disease and subsequent treatment, 2) the psychological effects of the disease and treatment, 3) the social, occupational, and financial impacts of the disease and treatment, 4) early detection of recurrence or subsequent primary malignancies, and last but not least, 5) prevention of cancer and promotion of healthy lifestyles.

The proposed questionnaire should effectively and comprehensively reflect both the physical problems typically associated with a given diagnosis and the psychological, social, occupational, and financial impacts. It should also focus the physician's attention on interventions aimed at healthy lifestyles (smoking cessation, obesity prevention, sufficient physical activity) to maintain the health of cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* The patient understands the information provided and agrees to participate in the study.
* Age 18 years or older.
* Histologically confirmed invasive breast cancer or invasive prostate cancer.
* Completion of the acute phase of curative oncological therapy:

  * for breast cancer: curative surgery performed + completed neoadjuvant/adjuvant chemotherapy and completed adjuvant radiotherapy, if indicated
  * for prostate cancer: completed radiotherapy with curative intent or radical prostatectomy performed (open, laparoscopic, robotic) or completed adjuvant radiotherapy after prostatectomy
* The patient is available for follow-up within 12 months of enrollment in the study.

Exclusion Criteria:

* Active ongoing oncological therapy (except for (i) adjuvant hormone therapy, (ii) adjuvant targeted therapy (anti-HER2 therapy, CDK4/6i, PARPi, T-DM1), (iii) adjuvant immunotherapy)
* Neoadjuvant/adjuvant therapy did not include chemotherapy (breast cancer).
* Recurrence of cancer
* Metastatic disease
* History of other primary malignancy (except for non-melanoma skin cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Impact of active monitoring of adverse effects on quality of life | Upon enrollment (baseline), six and twelve months after baseline
  Compare the quality of life of breast and prostate cancer survivors between the interventional group, in which adverse effects are actively monitored using the Questionnaire for the Assessment of Difficulties after Cancer Treatment, and the control group.

SECONDARY OUTCOMES:
Comprehensibility of the questionnaire | Upon enrollment (baseline), six and twelve months after baseline
  Evaluation of the comprehensibility of the Questionnaire for the Assessment of Difficulties after Cancer Treatment.
Usability of the questionnaire in routine clinical practice | Upon enrollment (baseline), six and twelve months after baseline
  Evaluation of the usability of the Questionnaire for the Assessment of Difficulties in routine clinical practice.
Frequency of active intervention by a physician | Upon enrollment (baseline), six and twelve months after baseline
  Assessment of the impact of active monitoring of adverse effects, based on the Questionnaire for the Assessment of Difficulties after Cancer Treatment, on the frequency of active physician interventions in the interventional group.

CONTACTS AND LOCATIONS:
Locations (1):
- Masaryk Memorial Cancer Institute, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Yes
IPD to be shared in pseudonymized form during the study. IPD to be published in anonymized form.
Supporting Information: CSR
Time Frame: after study completion
Access Criteria: During the study, data will be managed in pseudonymized form in a protected database environment, available only for study team.
  After completion of the study, the data will be fully anonymized for publication purposes. All publication outputs of the study will be carried out by a team of researchers led by the principal investigator. The submission of each publication is subject to the approval of the principal investigator.
  The results of this study may be published or presented at scientific meetings after approval by the PI and always after anonymization of the subjects' personal data in accordance with Act No. 101/2000 Coll., on the protection of personal data.
URL: https://www.mou.cz/veda-a-vyzkum/t1481

REFERENCES:
- [Background] Vaz-Luis I, Masiero M, Cavaletti G, Cervantes A, Chlebowski RT, Curigliano G, Felip E, Ferreira AR, Ganz PA, Hegarty J, Jeon J, Johansen C, Joly F, Jordan K, Koczwara B, Lagergren P, Lambertini M, Lenihan D, Linardou H, Loprinzi C, Partridge AH, Rauh S, Steindorf K, van der Graaf W, van de Poll-Franse L, Pentheroudakis G, Peters S, Pravettoni G. ESMO Expert Consensus Statements on Cancer Survivorship: promoting high-quality survivorship care and research in Europe. Ann Oncol. 2022 Nov;33(11):1119-1133. doi: 10.1016/j.annonc.2022.07.1941. Epub 2022 Aug 10. PMID 35963481
- [Background] Culbertson MG, Bennett K, Kelly CM, Sharp L, Cahir C. The psychosocial determinants of quality of life in breast cancer survivors: a scoping review. BMC Cancer. 2020 Oct 2;20(1):948. doi: 10.1186/s12885-020-07389-w. PMID 33008323
- [Background] van Leeuwen M, Kieffer JM, Efficace F, Fossa SD, Bolla M, Collette L, Colombel M, De Giorgi U, Holzner B, van de Poll-Franse LV, van Poppel H, White J, de Wit R, Osanto S, Aaronson NK; European Organisation for Research and Treatment of Cancer Quality of Life Group; Genito-Urinary Cancers Group and Radiation Oncology Group; and the NCRN Testis Clinical Studies Group. International evaluation of the psychometrics of health-related quality of life questionnaires for use among long-term survivors of testicular and prostate cancer. Health Qual Life Outcomes. 2017 May 11;15(1):97. doi: 10.1186/s12955-017-0670-4. PMID 28490338
- [Background] Allen I, Hassan H, Sofianopoulou E, Eccles D, Turnbull C, Tischkowitz M, Pharoah P, Antoniou AC. Risks of second non-breast primaries following breast cancer in women: a systematic review and meta-analysis. Breast Cancer Res. 2023 Feb 10;25(1):18. doi: 10.1186/s13058-023-01610-x. PMID 36765408
- [Background] Lustberg MB, Reinbolt RE, Shapiro CL. Bone health in adult cancer survivorship. J Clin Oncol. 2012 Oct 20;30(30):3665-74. doi: 10.1200/JCO.2012.42.2097. Epub 2012 Sep 24. PMID 23008309
- [Background] Mehta LS, Watson KE, Barac A, Beckie TM, Bittner V, Cruz-Flores S, Dent S, Kondapalli L, Ky B, Okwuosa T, Pina IL, Volgman AS; American Heart Association Cardiovascular Disease in Women and Special Populations Committee of the Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; and Council on Quality of Care and Outcomes Research. Cardiovascular Disease and Breast Cancer: Where These Entities Intersect: A Scientific Statement From the American Heart Association. Circulation. 2018 Feb 20;137(8):e30-e66. doi: 10.1161/CIR.0000000000000556. Epub 2018 Feb 1. PMID 29437116
- [Background] Nardin S, Mora E, Varughese FM, D'Avanzo F, Vachanaram AR, Rossi V, Saggia C, Rubinelli S, Gennari A. Breast Cancer Survivorship, Quality of Life, and Late Toxicities. Front Oncol. 2020 Jun 16;10:864. doi: 10.3389/fonc.2020.00864. eCollection 2020. PMID 32612947
- [Background] Mayer DK, Nasso SF, Earp JA. Defining cancer survivors, their needs, and perspectives on survivorship health care in the USA. Lancet Oncol. 2017 Jan;18(1):e11-e18. doi: 10.1016/S1470-2045(16)30573-3. PMID 28049573
- [Background] van Leeuwen M, Husson O, Alberti P, Arraras JI, Chinot OL, Costantini A, Darlington AS, Dirven L, Eichler M, Hammerlid EB, Holzner B, Johnson CD, Kontogianni M, Kjaer TK, Morag O, Nolte S, Nordin A, Pace A, Pinto M, Polz K, Ramage J, Reijneveld JC, Serpentini S, Tomaszewski KA, Vassiliou V, Verdonck-de Leeuw IM, Vistad I, Young TE, Aaronson NK, van de Poll-Franse LV; EORTC QLG. Understanding the quality of life (QOL) issues in survivors of cancer: towards the development of an EORTC QOL cancer survivorship questionnaire. Health Qual Life Outcomes. 2018 Jun 4;16(1):114. doi: 10.1186/s12955-018-0920-0. PMID 29866185
- See also: Institute of Health Information and Statistics of the Czech Republic — https://www.uzis.cz/index-en.php